CLINICAL TRIAL: NCT01270490
Title: A Multicentre, Prospective, Randomized Open-label Pilot Study to Assess the Feasibility and Preliminary Efficacy of Interferon-gamma in Combination With Anidulafungin for the Treatment of Candidemia
Brief Title: Efficacy of Interferon-gamma in Combination With Anidulafungin for the Treatment of Candidemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Principal Investigator, Corine Delsing, Drs, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interferon-gamma 001; 2009-014600-66 (EudraCT Number); NL28823.091.10 (Other: Dutch Central Committee on Research inv. Human Subjects)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Candidemia
Keywords: candidemia; candida sepsis; invasive fungal disease
MeSH Terms: conditions — Candidemia; Invasive Fungal Infections | interventions — Interferon-gamma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferon-gamma (Experimental)
  Interventions: Drug: Interferon-gamma, Recombinant
- No intervention (No Intervention): No adjunctive treatment

INTERVENTIONS:
Drug: Interferon-gamma, Recombinant — Interferon 50 mcg/m2 to be administered three times per week during two weeks
  Arms: Interferon-gamma

SUMMARY:
The purpose of this study is to assess the feasibility and preliminary efficacy of interferon-gamma in combination with anidulafungin for the treatment of candidemia

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females (who must agree to use barrier methods of contraception during the study therapy period, women of childbearing age must have a negative urine pregnancy or serum test at baseline).
* Subjects who are 18 years of age or older
* Subjects with at least one positive blood culture isolation of Candida species from a specimen drawn within 96 hours prior to study entry.
* Subjects who have clinical evidence of infection AT SOME TIME WITHIN 96 HOURS PRIOR TO ENROLLMENT, including AT LEAST ONE of the following:

  * Temperature >37.8 ˚C on 2 occasions at least 4 hours apart or one measurement > 38.2 ˚C
  * Systolic blood pressure <90 or a >30 mmHg decrease in systolic BP from the subject's normal baseline.
  * Signs of inflammation (swelling, heat, erythema, purulent drainage) from a site infected with Candida (eg, joint, skin, eye, bone, esophagus)
  * Radiologic findings of invasive candidiasis
* Subject or their legal representative must sign a written informed consent form.

Exclusion Criteria:

* Subjects with a history of allergy or intolerance to echinocandins or IFNgamma
* Subjects with a history of documented epileptic seizures
* Subjects with severe renal impairment (creatinine clearance less than 30/mL/min)
* Subjects with severe liver failure (impaired synthesis of proteins such as coagulation factors manifested by increased prothrombin time)
* Subjects with an absolute neutrophil count of less than 500/mm3 at study entry
* Women who are pregnant or lactating
* Subjects who are unlikely to survive more than 24 hours
* Subjects who have failed previous systemic antifungal therapy for the Candida spp. infection which is being studied.
* Subjects who have received more than 48 hours of systemic antifungal therapy for the current episode, within 96 hours prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
the time to negative blood cultures | at fixed time points during follow up (at least until 8 weeks after end of treatment)

SECONDARY OUTCOMES:
overall survival | until 8 weeks after end of treatment
time to death | Until 8 weeks after end of treatment
outcome of fungal infection | Until 8 weeks after end of treatment
  resolution at week 2 and 8 after end of treatment, patient status at end of therapy, microbiological parameters
duration of antifungal therapy | Until end of treatment
duration of hospitalization | Until end of hospitilization
immunological parameters | Until 8 weeks after end of treatment
tolerability and safety | until 8 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Netea, MD PhD, Study Director — Radboud University Medical Center; Corine Delsing, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Derived] Delsing CE, Gresnigt MS, Leentjens J, Preijers F, Frager FA, Kox M, Monneret G, Venet F, Bleeker-Rovers CP, van de Veerdonk FL, Pickkers P, Pachot A, Kullberg BJ, Netea MG. Interferon-gamma as adjunctive immunotherapy for invasive fungal infections: a case series. BMC Infect Dis. 2014 Mar 26;14:166. doi: 10.1186/1471-2334-14-166. PMID 24669841